CLINICAL TRIAL: NCT01649908
Title: Evaluation of Cardiac Function in Different Techniques in Infrarenal Aortic Surgery
Brief Title: Open Bifurcation Surgery Study
Acronym: OBI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alexander Hyhlik-Duerr, M. D. (Other)
Collaborators: Vascutek Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Alexander Hyhlik-Duerr, M. D., M.D., Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: 501961
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Infrarenal Aortic Aneurysm

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- sectional cross clamping
- simultaniously cross clamping
- EVAR

SUMMARY:
Different cross clamping techniques in aortic surgery causes different cardiac stress

ELIGIBILITY:
Inclusion Criteria:

* AAA > 5cm

Exclusion Criteria:

* emergency cases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infrarenal aortic aneurysms
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-07

PRIMARY OUTCOMES:
cardiac function with echocardiography | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- See also: Related Info — http://www.klinikum.uni-heidelberg.de/Home.104613.0.html